CLINICAL TRIAL: NCT00613366
Title: Effect of Prophylactic Misoprostol Prior to Intrauterine Device Insertion
Brief Title: Misoprostol With Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, MD MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OHSU RES 3489
Record Dates: First submitted 2008-01-29; First posted 2008-02-13 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-02

CONDITIONS: Contraception
Keywords: intrauterine device; cervical dilation; nulliparous women; pain management
MeSH Terms: conditions — Agnosia | interventions — Misoprostol; Prostaglandins; Magnesium Oxide; Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): Cervical preparation with misoprostol prior to intrauterine device insertion
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Cervical preparation with placebo prior to intrauterine device insertion
  Interventions: Dietary Supplement: Magnesium Oxide

INTERVENTIONS:
Drug: Misoprostol — Place 2 tablets between the teeth and cheek and allow to dissolve for 30 minutes.
  Other Names: prostaglandin
  Arms: Misoprostol
Dietary Supplement: Magnesium Oxide — Place 2 tablets between the teeth and cheek and allow to dissolve for 30 minutes.
  Other Names: Magnesium; Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if using misoprostol (a medication that softens the cervix) before placing an intrauterine device for contraception reduces pain in women who have never delivered a baby.

DETAILED DESCRIPTION:
The investigators intend to conduct a randomized double blind study at Oregon Health and Science University and Planned Parenthood of the Columbia Willamette.

Subjects will be approached only after deciding to get an intrauterine. When the participants return for intrauterine device placement, at 90 minutes prior to the procedure half will receive misoprostol and half will receive placebo. The subjects will be asked to rate their level of pain at specific points during the insertion. Providers will be asked to mark whether or not additional dilation was required as well as their perceived ease of intrauterine device placement.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women (defined as those without a history of pregnancy, despite the outcome, beyond 20 weeks gestation)
* Ages 18-45
* Seeking long-term reversible contraception with an intrauterine device (either Mirena or Paraguard) through the OHSU Center for Women's Health and Planned Parenthood of the Columbia Willamette

Exclusion Criteria:

* Pregnancy occurring less than 6 weeks from time of presentation
* History of prior intrauterine device placement
* History of Mullerian tract anomalies
* History of uterine surgery
* Allergy or intolerance to misoprostol or other prostaglandin
* Pelvic inflammatory disease (current or within the past 3 months)
* Sexually transmitted diseases (current)
* Puerperal or postabortion sepsis (current or within the past 3 months)
* Purulent cervicitis (current)
* Undiagnosed abnormal vaginal bleeding
* Malignancy of the genital tract
* Known uterine anomalies or fibroids distorting the cavity in a way incompatible with intrauterine device insertion
* Allergy to any component of the intrauterine device or Wilson's disease (for copper- containing intrauterine device)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, M.D., M.P.H, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Planned Parenthood of the Columbia Willamette, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Derived] Turok DK, Espey E, Edelman AB, Lotke PS, Lathrop EH, Teal SB, Jacobson JC, Simonsen SE, Schulz KF. The methodology for developing a prospective meta-analysis in the family planning community. Trials. 2011 Apr 29;12:104. doi: 10.1186/1745-6215-12-104. PMID 21527040
- See also: (Women's Health Research Unit website) — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2007-March 2010 in general OB/GYN clinic at an academic hospital
Pre-assignment Details: Women desiring IUD placement who were nulliparous were enrolled.
Groups:
- Active Drug (Misoprostol): 400mcg of buccal misoprostol 90 minutes prior to IUD insertion
- Placebo: Placebo buccal 90 minutes prior to IUD insertion.
Period: Overall Study
Arm/Group | Active Drug (Misoprostol) | Placebo
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug (Misoprostol) | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 27 (6) | 26 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: The Ease of IUD Insertion as Rated by the Provider Using a 100mm Visual Analog Scale (VAS).
Description: Provider ease of insertion was measured using a 100mm visual analog scale (VAS).The 100mm Pain Visual Analog Scale (VAS) is an instrument used to capture subjective attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of pain by indicating a position along a 100mm continues line: pain scores can range from 0="No Pain" (furthest point to the left) to 100="Worst Pain of My Life" (furthest point to the right).
Time Frame: Time of IUD insertion
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active Drug (Misoprostol) | Placebo
Number analyzed (Participants) | 17 | 18
mm | 24 (19) | 29 (21)

2. Secondary Outcome: Perceived Pain of IUD Insertion by Patient Using a 100mm Visual Analog Scale (VAS).
Description: Perceived pain measured using a 100mm visual analog scale (VAS).The 100mm Pain Visual Analog Scale (VAS) is an instrument used to capture subjective attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of pain by indicating a position along a 100mm continues line: pain scores can range from 0="No Pain" (furthest point to the left) to 100="Worst Pain of My Life" (furthest point to the right).
Time Frame: At time of IUD insertion
Population: ITT
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active Drug (Misoprostol) | Placebo
Number analyzed (Participants) | 17 | 18
mm | 65 (21) | 55 (21)

ADVERSE EVENTS:
Arm/Group | Active Drug (Misoprostol) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No